CLINICAL TRIAL: NCT00185276
Title: Randomized, Multi-center Open Label Study of the Safety (Open-label) and Efficacy (Open-label & Blinded Reader) of Magnevist® Injection-enhanced Magnetic Resonance Arteriography (MRA) at Two Dose Levels and 2-dimensional-time-of-flight (2D-TOF) MRA in Patients Undergoing MRA of the Infrarenal Aorta and Peripheral Arteries With Intra-arterial Digital Subtraction Arteriography (i.a. DSA) as Standard of Reference
Brief Title: Magnevist® Injection Enhanced MRA at Two Dose Levels Compared to Non Contrast MRA for the Detection of Structural Abnormalities of the Infrarenal Aorta and Peripheral Arteries
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 91208; 306781
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Peripheral Vascular Disease
Keywords: Structural abnormalities of the infrarenal aorta and peripheral arteries
MeSH Terms: conditions — Peripheral Vascular Diseases | interventions — Gadolinium DTPA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Gadopentetate dimeglumine (Magnevist, BAY86-4882)
- Arm 2 (Experimental)
  Interventions: Drug: Gadopentetate dimeglumine (Magnevist, BAY86-4882)

INTERVENTIONS:
Drug: Gadopentetate dimeglumine (Magnevist, BAY86-4882) — Single intravenous injection on the study day: lower dose corresponding approx. 0.1 mmol/kg body weight
  Arms: Arm 1
Drug: Gadopentetate dimeglumine (Magnevist, BAY86-4882) — Single intravenous injection on the study day: higher dose corresponding approx. 0.2 - 0.3 mmol/kg body weight
  Arms: Arm 2

SUMMARY:
The purpose of this study is to look at the safety (what are the side effects) and efficacy (how well does it work) of Magnevist (the study drug) used for MRI of the infrarenal aorta and peripheral arteries. The results will be compared to the results of MRI taken without Magnevist, and with the results of your X-ray angiography.

DETAILED DESCRIPTION:
This study has previously been posted by Berlex, Inc. Berlex, Inc. has been renamed to Bayer HealthCare Pharmaceuticals, Inc.Bayer HealthCare Pharmaceuticals, Inc.is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Has known or suspected peripheral vascular disease
* Is scheduled for X-ray angiography

Exclusion Criteria:

* Has any contraindication to magnetic resonance imaging
* Is scheduled for any procedure before the X-ray angiography
* Had previously had stents placed bilaterally in the region to be imaged

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2003-03; Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Sensitivity, specificity and accuracy of the higher dose of Magnevist® Injection and 2D-TOF MRA for the detection of clinically significant disease | Image creation after injection - evaluation at blind read

SECONDARY OUTCOMES:
Diagnostic confidence | At blinded or/and open label read of images
Visual assessment of stenosis | At blinded or/and open label read of images
Difference in degree of stenosis | At blinded or/and open label read of images
Other diagnostic findings | At blinded or/and open label read of images
Image quality | At blinded or/and open label read of images
Image evaluability and presence of artifacts | At blinded or/and open label read of images
Ability to visualize arterial segments | At blinded or/and open label read of images
Number of evaluable segments | At blinded or/and open label read of images
Location and matching of stenosis | At blinded or/and open label read of images
SI measurements | At blinded or/and open label read of images
Patient management | From baseline to 24 hours follow-up
Safety | From baseline to 24 hours follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer